CLINICAL TRIAL: NCT03334435
Title: A Phase 3 Multicenter, Double-Blind Study to Evaluate the Long-Term Safety and Efficacy of Baricitinib in Adult Patients With Atopic Dermatitis
Brief Title: A Study of Long-term Baricitinib (LY3009104) Therapy in Atopic Dermatitis
Acronym: BREEZE-AD3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16587; I4V-MC-JAHN (Other: Eli Lilly and Company); 2017-000873-35 (EudraCT Number)
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2022-07-01 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Responders and Partial Responders (RPR)-Placebo (Placebo Comparator): Responders or partial responders (RPR) [Investigator's Global Assessment (IGA) of (0,1, or 2) at entry to study JAHN and never rescued in originating study] participants from previous Baricitinib monotherapy studies-JAHL and JAHM and combination therapy study-JAIY were assigned to remain in this arm to receive placebo orally.
  Interventions: Drug: Baricitinib; Drug: Placebo
- RPR-Bari 1-milligram (mg) (Experimental): RPR participants from previous Baricitinib monotherapy studies-JAHL and JAHM were assigned to remain in this arm to receive Baricitinib 1 mg orally.
  Interventions: Drug: Baricitinib
- RPR-Bari 2-mg (Experimental): RPR participants from previous Baricitinib monotherapy studies-JAHL and JAHM and combination therapy study-JAIY were assigned to remain in this arm to receive Baricitinib 2 mg orally.
  Interventions: Drug: Baricitinib
- RPR-Bari 4-mg (Experimental): RPR participants from previous Baricitinib monotherapy studies-JAHL and JAHM and combination therapy study-JAIY were assigned to remain in this arm to receive Baricitinib 4 mg orally.
  Interventions: Drug: Baricitinib
- Non-responders (NR): Bari 1 mg to 2 mg (Experimental): Non-responder (NR) [those not meeting definition of RPR] participants from previous Baricitinib monotherapy studies-JAHL and JAHM who received Baricitinib 1 mg and were re-randomized to this arm to receive Baricitinib 2 mg orally.
  Interventions: Drug: Baricitinib
- NR: Bari 1 mg to 4 mg (Experimental): NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM who received Baricitinib 1 mg and were re-randomized to this arm to receive Baricitinib 4 mg orally.
  Interventions: Drug: Baricitinib
- NR: Bari 2 mg to 2 mg (Experimental): NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM and combination therapy study-JAIY who received Baricitinib 2 mg and were re-randomized to this arm to receive Baricitinib 2 mg orally.
  Interventions: Drug: Baricitinib
- NR: Bari 2 mg to 4 mg (Experimental): NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM and combination therapy study-JAIY who received Baricitinib 2 mg and were re-randomized to this arm to receive Baricitinib 4 mg orally.
  Interventions: Drug: Baricitinib
- NR: Bari 4 mg to 4 mg (Experimental): NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM and combination therapy study-JAIY who received Baricitinib 4 mg and were re-randomized to this arm to receive Baricitinib 4 mg orally.
  Interventions: Drug: Baricitinib
- NR: Placebo to Bari 2 mg (Experimental): NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM and combination therapy study-JAIY who received placebo and were re-randomized to this arm to receive Baricitinib 2 mg orally.
  Interventions: Drug: Baricitinib; Drug: Placebo
- NR: Placebo to Bari 4 mg (Experimental): NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM and combination therapy study-JAIY who received placebo and were re-randomized to this arm to receive Baricitinib 4 mg orally.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo (Placebo Comparator): Participants from previous Baricitinib monotherapy studies (JAHL, JAHM) and combination therapy study (JAIY) were randomized or assigned to this arm to receive placebo orally.
  Interventions: Drug: Placebo
- Bari 1 mg (Experimental): Participants from previous Baricitinib monotherapy studies (JAHL, JAHM) were randomized or assigned to this arm to receive Baricitinib 1 mg orally.
  Interventions: Drug: Baricitinib
- Bari 2 mg (Experimental): Participants from previous Baricitinib monotherapy studies (JAHL, JAHM) and combination therapy study (JAIY) were randomized or assigned to this arm to receive Baricitinib 2 mg orally.
  Interventions: Drug: Baricitinib
- Bari 4 mg (Experimental): Participants from previous Baricitinib monotherapy studies (JAHL, JAHM) and combination therapy study (JAIY) were randomized or assigned to this arm to receive Baricitinib 4 mg orally.
  Interventions: Drug: Baricitinib
- Bari 2-mg Open-Label Addendum (Experimental): Participants were directly enrolled to this open-label arm to receive Baricitinib 2-mg orally.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: Bari 1 mg; Bari 2 mg; Bari 2-mg Open-Label Addendum; Bari 4 mg; NR: Bari 1 mg to 4 mg; NR: Bari 2 mg to 2 mg; NR: Bari 2 mg to 4 mg; NR: Bari 4 mg to 4 mg; NR: Placebo to Bari 2 mg; NR: Placebo to Bari 4 mg; Non-responders (NR): Bari 1 mg to 2 mg; RPR-Bari 1-milligram (mg); RPR-Bari 2-mg; RPR-Bari 4-mg; Responders and Partial Responders (RPR)-Placebo
Drug: Placebo — Administered orally
  Arms: NR: Placebo to Bari 2 mg; NR: Placebo to Bari 4 mg; Placebo; Responders and Partial Responders (RPR)-Placebo

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of baricitinib in participants with atopic dermatitis.

Participants were enrolled in this study from the originating studies (JAHL, JAHM, JAIY) or were directly enrolled in the open-label arm.

ELIGIBILITY:
Have participated in previous studies (JAHL, JAHM and JAIY) and met specific completion requirements for those studies, and do not meet any of the following Exclusions:

Exclusion Criteria:

* Had investigational product permanently discontinued at any time during a previous Baricitinib study.
* Had temporary investigational product interruption continue at the final study visit of a previous Baricitinib study and, in the opinion of the investigator, this poses an unacceptable risk for the participant's participation in the study

OR

Have not participated in previous studies (JAHL, JAHM and JAIY) and satisfy the following criteria:

Inclusion Criteria:

* Have been diagnosed with moderate to severe Atopic Dermatitis for at least 12 months.
* Have had inadequate response or intolerance to existing topical (applied to the skin) medications within 6 months preceding screening.
* Are willing to discontinue certain treatments for eczema (such as systemic and topical treatments during a washout period).
* Agree to use emollients daily.

Exclusion Criteria:

* Are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus), or a history of erythrodermic, refractory, or unstable skin disease that requires frequent hospitalizations and/or intravenous treatment for skin infections.
* A history of eczema herpeticum within 12 months, and/or a history of 2 or more episode of eczema herpeticum in the past.
* Participants who are currently experiencing a skin infection that requires treatment, or is currently being treated, with topical or systemic antibiotics.
* Have any serious illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g., unstable chronic asthma).
* Have been treated with the following therapies:

  * Monoclonal antibody for less than 5 half-lives prior to randomization.
  * Received prior treatment with any oral Janus kinase (JAK) inhibitor.
  * Received any parenteral corticosteroids administered by intramuscular or intravenous (IV) injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization or are anticipated to require parenteral injection of corticosteroids during the study.
  * Have had an intra-articular corticosteroid injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization.
* Have high blood pressure characterized by a repeated systolic blood pressure >160 millimeters of mercury (mm Hg) or diastolic blood pressure >100 mm Hg.
* Have had major surgery within the past eight weeks or are planning major surgery during the study.
* Have experienced any of the following within 12 weeks of screening: venous thromboembolic event (VTE), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have a history of recurrent (≥ 2) VTE or are considered at high risk of VTE as deemed by the investigator.
* Have a history or presence of cardiovascular, respiratory, hepatic, chronic liver disease gastrointestinal, endocrine, hematological, neurological, lymphoproliferative disease or neuropsychiatric disorders or any other serious and/or unstable illness.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection including herpes zoster, tuberculosis.
* Have specific laboratory abnormalities.
* Have received certain treatments that are contraindicated.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1645 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (185):
- Argentina (7):
  - CEDIC-Centro de Investigaciones Clinicas, Caba, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Buenos Aires Skin, Ciudad Autonoma Buenos Aires
  - Fundacion CIDEA, Ciudad Autonoma Buenos Aires
  - Instituto de Neumonología y Dermatología, Ciudad Autonoma Buenos Aires
  - Psoriahue Medicina Interdisciplinaria, Ciudad Autonoma Buenos Aires
  - Parra Dermatología, Mendoza
- Australia (7):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Skin & Cancer Foundation Australia, Westmead, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Clinical Trials SA Pty Ltd, Adelaide, South Australia
  - Skin and Cancer Foundation Inc., Carlton, Victoria
  - Fremantle Dermatology, Perth, Western Australia
- Austria (6):
  - Universitätsklinikum Graz, Graz, Styria
  - Ordensklinikum Linz GmbH - Elisabethinen, Linz, Upper Austria
  - KA Rudolfstiftung, Vienna
  - AKH, Vienna
  - KH Hietzing mit neurologischem Zentrum Rosenhügel, Vienna
  - Sozialmed. Zentrum Ost - Donauspital, Vienna
- Czechia (9):
  - Kozni ambulance Kutna Hora, s.r.o., Kutná Hora, Central Bohemia
  - Clintrial, s.r.o., Prague, Hl. M. Praha
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Hl. M. Praha
  - Fakultni Nemocnice v Motole, Prague, Hl. M. Praha
  - Nemocnice Na Bulovce, Prague, Hl. M. Praha
  - Nemocnice Novy Jicin a.s., Nový Jičín, Moravskoslezský kraj
  - Fakultni Nemocnice Plzen, Plzen-Bory, Plzeň Region
  - Fakultni Nemocnice U svate Anny, Brno, South Moravian
  - Krajska zdravotni a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem, Ustecký Kraj
- Denmark (2):
  - Gentofte Hospital, Hellerup, Capital Region
  - Aarhus Universitehospital Marselisborg Centret, Aarhus, Region Midtjyland
- France (7):
  - Hopital Saint-Louis, Paris, Cedex 10
  - CHU de Bordeaux Hopital Saint Andre, Bordeaux
  - CHU Grenoble Alpes, Grenoble Cédex 9
  - Chru De Nantes Hotel-Dieu, Nantes
  - CHU de Nice Hopital de L'Archet, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Larrey, Toulouse
- Germany (22):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum der Universität München, München, Bavaria
  - Gemeinschaftspraxis Mahlow, Blankenfelde-Mahlow, Brandenburg
  - Rosenpark Research Geschäftsbereich der Rosenparkklinik GmbH, Darmstadt, Hesse
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Dermatologisches Zentrum Osnabrück Nord, Bramsche, Lower Saxony
  - Universitätsmedizin Göttingen, Göttingen, Lower Saxony
  - Universitätsmedizin Rostock, Rostock, Mecklenburg-Vorpommern
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Praxis Gerlach, Dresden, Saxony
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universität Leipzig - Universitätsklinikum, Leipzig, Saxony
  - Universitätsklinikum Otto-von-Guericke-Universität, Magdeburg, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Universitätsklinikum Aachen AöR - Klinik für Dermatologie und Allergologie - Hautklinik, Aachen
  - Charité Universitätsmedizin Berlin, Berlin
  - Rothhaar Studien GmbH, Berlin
  - ISA GmbH, Berlin
  - Praxis für Ganzheitliche Dermatologie im Ärztehaus, Berlin
  - TFS Trial Form Support GmbH, Hamburg
- Hungary (9):
  - Oroshaza Varosi Onkormanyzat Korhaza, Orosháza, Bekes County
  - SZTE AOK Borgyogyaszati es Allergologiai Klinika, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont Borgyogyaszati Klinika, Debrecen, Hajdú-Bihar
  - Trial Pharma Kft., Püspökladány, Hajdú-Bihar
  - Allergo-Derm Bakos Kft, Szolnok, Jász-Nagykun-Szolnok
  - Kaposi Mor Oktato Korhaz, Kaposvár, Somogy County
  - Markusovszky Korhaz, Szombathely, Vas County
  - UNO Medical Trials Kft., Budapest
  - MedMare Bt, Veszprém
- India (8):
  - King George Hospital, Vizag, Andhra Pradesh
  - Panchshil Hospital, Ahmedabad, Gujarat
  - Byramjee Jeejeebhoy Medical College & Civil Hospital, Ahmedabad, Gujarat
  - Dr. D. Y. Patil Medical College & Hospital, Navi Mumbai, Maharashtra
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharshtra
  - All India Institue of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Gandhi Hospital, Secunderabad, Telangana
- Israel (6):
  - Haemek Medical Center- Dermatology, Afula
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Policlinico Univ. Agostino Gemelli, Rome, Lazio
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Universitaria Ospedale San Martino di Genova, Genova
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera - Universitaria Pisana, Pisa
  - Policlinico di Tor Vergata, Roma
  - Ospedale Policlinico Giambattista Rossi, Borgo Roma, Verona
  - ULSS 8, Vicenza
- Japan (36):
  - Yanagihara dermatology clinic, Ainokawa, Ichikawa-shi, Chiba
  - Kawashima Dermatology Clinic, Ichikawa-shi, Chiba
  - Medical Corporation Soleil Miyata Dermatology Clinic, Matsudo-shi, Chiba
  - Fumimori Clinic, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Shibaki Dermatology Clinic, Sapporo, Hokkaido
  - Sapporo Skin Clinic, Sapporo, Hokkaido
  - Tokyo Medical University Ibaraki Medical Center, Inashiki-gun, Ibaraki
  - Queen's Square Dermatology and Allergology, Nishi-ku, Yokohama-city, Kanagawa
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Noguchi Dermatology, Kashima-machi, Kamimashiki-gun, Kumamoto
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Kume Clinic, Nishi-ku Sakai-shi, Osaka
  - Senri-Chuo Hanafusa Dermatology Clinic, Toyonaka-shi, Osaka
  - Sanrui Dermatology Clinic, Ohmiya-ku,Saitama-shi, Saitama
  - Shimane University Hospital, Izumo, Shimane
  - JA Shizuoka Kohseiren Enshu Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Iidabashi Clinic, Chiyoda-ku, Tokyo
  - Tokyo Teishin Hospital, Chiyoda-Ku, Tokyo
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Hosono Clinic, Chuo-ku, Tokyo
  - Sumire Dermatology Clinic, Edogawa-ku, Tokyo
  - Oizumi Hanawa Clinic, Nerima-ku, Tokyo
  - Naoko Dermatology Clinic, Setagaya-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-KU, Tokyo
  - Yamate Dermatological Clinic, Shinjuku, Tokyo
  - Tachikawa Dermatology Clinic, Tachikawa-shi, Tokyo
  - Shirasaki Clinic, Takaoka-shi, Toyama
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Gifu University Hospital, Gifu
  - Osaka City University Hospital, Osaka
- Mexico (8):
  - Grupo Medico Camino S.C., Mexico City, Mexico City
  - Hospital de Jesus I.A.P., Mexico City, Mexico City
  - Clinica De Enfermedades Cronicas y Procedimientos Especiales, Morelia, Michoacan Morelia
  - CRI Centro Regiomontano de Investigacion S.C., Monterrey, Nuevo León
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - JM Research S.C., Cuernavaca
  - RM Pharma Specialists S.A. de C.V., Distrito Federal
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C, Durango
- Poland (13):
  - DermoDent, Centrum Medyczne Czajkowscy, Osielsko, Kuyavian-Pomeranian Voivodeship
  - Barbara Rewerska DIAMOND CLINIC, Krakow, Lesser Poland Voivodeship
  - Lubelskie Centrum Diagnostyczne, Świdnik, Lublin Voivodeship
  - Centrum Medyczne AMED, Warsaw, Masovian Voivodeship
  - Centralny Szpital Kliniczny MSWiA, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Evimed, Warsaw, Masovian Voivodeship
  - Wojskowy Instytut Medyczny CSK MON, Warsaw, Masovian Voivodeship
  - NZOZ Specjalistyczna Przychodnia Dermatologiczna Specderm, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych, PI House, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Miejski Szpital Zespolony w Olsztynie Klinika Dermatologii, Olsztyn, Warmian-Masurian Voivodeship
  - LASER CLINIC Specjalistyczne Gabinety Lekarskie, Szczecin, West Pomeranian Voivodeship
  - Dermed Centrum Medyczne Sp. z o.o., Lodz, Łódź Voivodeship
- Russia (6):
  - GBUZ Clinical dermatology and venereological dispensary, Krasnodar, Krasnodarskiy Kray
  - State scientific centre for dermatovenerology and cosmetolog, Moscow
  - Russian state medical-stomatological university n.a. Evdokimov, Moscow
  - SPb SBHI Skin-venerologic dispensary #10, Saint Petersburg
  - LLC ArsVitae NorthWest, Saint Petersburg
  - LLC Medical Center "Kurator", Saint Petersburg
- South Korea (9):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Korea
  - Severance Hospital Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Chungang University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (11):
  - Hospital Germans Trias i Pujol, Barcelona, Badalona
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Clinica Universitaria De Navarra, Pamplona, Navarre
  - Hospital General Universitario Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital De Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro de Especialidades Mollabao, Pontevedra
- Switzerland (4):
  - CHUV Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Inselspital Bern, Bern
  - HUG-Hôpitaux Universitaires de Genève, Geneva
  - Universitätsspital Zürich, Zurich
- Taiwan (7):
  - Chang Gung Memorial Hospital - Linkou, Taoyuan, (r.o.c.), Taiwan
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Taipei Medical University- Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Taipei, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- [Derived] Thyssen JP, Werfel T, Barbarot S, Hunter HJA, Pierce E, Sun L, Cirri L, Buchanan AS, Lu N, Wollenberg A. Maintained improvement in physician- and patient-reported outcomes with baricitinib in adults with moderate-to-severe atopic dermatitis who were treated for up to 104 weeks in a randomized trial. J Dermatolog Treat. 2023 Dec;34(1):2190430. doi: 10.1080/09546634.2023.2190430. PMID 36912484
- [Derived] Reich K, Simpson E, Wollenberg A, Bissonnette R, Abe M, Cardillo T, Janes J, Sun L, Chen S, Silverberg JI. Efficacy of downtitration or treatment withdrawal compared with continuous dosing after successful treatment with baricitinib in patients with moderate-to-severe atopic dermatitis in a randomized substudy from the long-term extension study BREEZE-AD3. Br J Dermatol. 2023 Feb 10;188(2):208-217. doi: 10.1093/bjd/ljac057. PMID 36763879
- [Derived] Wollenberg A, Kircik L, Simpson E, Brinker D, Katoh N, Rueda MJ, Issa M, Yang F, Feely M, Alexis A. Pooled Analysis of Baricitinib Tolerability in Patients With Atopic Dermatitis in Relation to Acne, Headache, and Gastrointestinal Events From 8 Clinical Trials. Dermatitis. 2023 Jul-Aug;34(4):308-314. doi: 10.1089/derm.2022.0027. Epub 2023 Feb 6. PMID 36749121
- [Derived] Katoh N, Takita Y, Isaka Y, Nishikawa A, Torisu-Itakura H, Saeki H. Pooled Safety Analysis of Baricitinib in Adult Participants with Atopic Dermatitis in the Japanese Subpopulation from Six Randomized Clinical Trials. Dermatol Ther (Heidelb). 2022 Dec;12(12):2765-2779. doi: 10.1007/s13555-022-00828-5. Epub 2022 Oct 18. PMID 36255569
- [Derived] Silverberg JI, Simpson EL, Wollenberg A, Bissonnette R, Kabashima K, DeLozier AM, Sun L, Cardillo T, Nunes FP, Reich K. Long-term Efficacy of Baricitinib in Adults With Moderate to Severe Atopic Dermatitis Who Were Treatment Responders or Partial Responders: An Extension Study of 2 Randomized Clinical Trials. JAMA Dermatol. 2021 Jun 1;157(6):691-699. doi: 10.1001/jamadermatol.2021.1273. PMID 33978711
- [Derived] King B, Maari C, Lain E, Silverberg JI, Issa M, Holzwarth K, Brinker D, Cardillo T, Nunes FP, Simpson EL. Extended Safety Analysis of Baricitinib 2 mg in Adult Patients with Atopic Dermatitis: An Integrated Analysis from Eight Randomized Clinical Trials. Am J Clin Dermatol. 2021 May;22(3):395-405. doi: 10.1007/s40257-021-00602-x. Epub 2021 Apr 7. PMID 33826132
- See also: A Study of Long-term Baricitinib (LY3009104) Therapy in Atopic Dermatitis (Eczema) (BREEZE-AD3) — https://trials.lillytrialguide.com/en-US/trial/64kocErmNim2YSiiqCaOk6

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who entered Study JAHN were classified as "Responders and Partial Responders (RPR): Investigator's Global Assessment (IGA) of (0, 1, or 2) at entry to study JAHN and never rescued in originating study" or "Non-responders (NR): those not meeting definition of RPR". The study has two treatment periods: Treatment period 1, from Week 0 up to Week 52, and Treatment period 2, from Week 52 through Week 200 which included randomized withdrawal and downtitration substudy (RWDT).
Groups:
- Baricitinib (Bari) 1- Milligram (mg): Participants from previous Baricitinib monotherapy studies (JAHL, JAHM) were randomized or assigned to this arm to receive Baricitinib 1 mg orally.
- Bari 2-mg: Participants from previous Baricitinib monotherapy studies (JAHL, JAHM) and combination study (JAIY) were randomized or assigned to this arm to receive Baricitinib 2 mg orally.
- Bari 4-mg: Participants from previous Baricitinib monotherapy studies (JAHL, JAHM) and combination study (JAIY) were randomized or assigned to this arm to receive Baricitinib 4 mg orally.
- 2 mg Bari to Placebo Substudy: Participants who received Baricitinib 2 mg at the start of Study JAHN were rerandomized at week 52 or assigned to this arm to receive placebo orally.
- 2 mg Bari to 1 mg Bari Substudy: Participants who received Baricitinib 2 mg at the start of Study JAHN were rerandomized at week 52 or assigned to this arm to receive Baricitinib 1 mg orally.
- 2 mg Bari to 2 mg Bari Substudy: Participants who received Baricitinib 2 mg at the start of Study JAHN were rerandomized at week 52 or assigned to this arm to receive Baricitinib 2 mg orally.
- 4 mg Bari to Placebo Substudy: Participants who received Baricitinib 4 mg at the start of Study JAHN were rerandomized at week 52 or assigned to this arm to receive placebo orally.
- 4 mg Bari to 2 mg Bari Substudy: Participants who received Baricitinib 4 mg at the start of Study JAHN were rerandomized at week 52 or assigned to this arm to receive Baricitinib 2 mg orally.
- 4 mg Bari to 4 mg Bari Substudy: Participants who received Baricitinib 4 mg at the start of Study JAHN were rerandomized at week 52 or assigned to this arm to receive Baricitinib 4 mg orally.
- Placebo to Placebo Non-substudy: Participants who received placebo at the start of Study JAHN who were not eligible to enter the substudy at week 52 assigned to this arm to receive placebo orally.
- 1 mg Bari to 1 mg Bari Non-substudy: Participants who received Baricitinib 1 mg at the start of Study JAHN who were not eligible to enter the substudy at week 52 assigned to this arm to receive Baricitinib 1 mg orally.
- 2 mg Bari to 2 mg Bari Non-substudy: Participants who received Baricitinib 2 mg at the start of Study JAHN who were not eligible to enter the substudy at week 52 assigned to this arm to receive Baricitinib 2 mg orally.
- 4 mg Bari to 4 mg Bari Non-substudy: Participants who received Baricitinib 4 mg at the start of Study JAHN who were not eligible to enter the substudy at week 52 assigned to this arm to receive Baricitinib 4 mg orally.
Period: Treatment Period 1: Week 0 to Week 52
Arm/Group | Placebo | Baricitinib (Bari) 1- Milligram (mg) | Bari 2-mg | Bari 4-mg | Bari 2-mg Open-Label Addendum | 2 mg Bari to Placebo Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to 4 mg Bari Substudy | Placebo to Placebo Non-substudy | 1 mg Bari to 1 mg Bari Non-substudy | 2 mg Bari to 2 mg Bari Non-substudy | 4 mg Bari to 4 mg Bari Non-substudy
Started | 91 | 45 | 519 | 743 | 247 (Participants from the Bari 2-mg Open-Label Addendum were randomized into Treatment Period 2.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Investigational Product (IP) | 91 | 45 | 519 | 743 | 247 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RPR | 91 | 45 | 108 | 134 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NR | 0 | 0 | 411 | 609 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 12 | 15 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 89 | 43 | 507 | 728 | 242 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ongoing as of Week 52 (Later participants were moved to treatment period 2 [week 52 to 200]) | 70 | 32 | 379 | 519 | 146 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 5 | 76 | 140 | 61 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 9 | 23 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 4 | 38 | 42 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2: Week 52 to Week 200
Arm/Group | Placebo | Baricitinib (Bari) 1- Milligram (mg) | Bari 2-mg | Bari 4-mg | Bari 2-mg Open-Label Addendum | 2 mg Bari to Placebo Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to 4 mg Bari Substudy | Placebo to Placebo Non-substudy | 1 mg Bari to 1 mg Bari Non-substudy | 2 mg Bari to 2 mg Bari Non-substudy | 4 mg Bari to 4 mg Bari Non-substudy
Started | 0 (Participants were assigned to this arm only during treatment period 1,) | 0 (Participants were assigned to this arm only during treatment period 1,) | 0 (Participants were assigned to this arm only during treatment period 1,) | 0 (Participants were assigned to this arm only during treatment period 1,) | 0 (Participants were assigned to this arm only during treatment period 1,) | 92 (At Week 52: participants (with IGA 0, 1, or 2) who were assigned to Baricitinib 4 mg or 2 mg, at randomization were receiving IP and had not used high-potency TCS in the previous 14 days were enrolled in the RWDT substudy.) | 91 (At Week 52: participants (with IGA 0, 1, or 2) who were assigned to Baricitinib 4 mg or 2 mg, at randomization were receiving IP and had not used high-potency TCS in the previous 14 days were enrolled in the RWDT substudy.) | 92 (At Week 52: participants (with IGA 0, 1, or 2) who were assigned to Baricitinib 4 mg or 2 mg, at randomization were receiving IP and had not used high-potency TCS in the previous 14 days were enrolled in the RWDT substudy.) | 84 (At Week 52: participants (with IGA 0, 1, or 2) who were assigned to Baricitinib 4 mg or 2 mg, at randomization were receiving IP and had not used high-potency TCS in the previous 14 days were enrolled in the RWDT substudy.) | 84 (At Week 52: participants (with IGA 0, 1, or 2) who were assigned to Baricitinib 4 mg or 2 mg, at randomization were receiving IP and had not used high-potency TCS in the previous 14 days were enrolled in the RWDT substudy.) | 84 (At Week 52: participants (with IGA 0, 1, or 2) who were assigned to Baricitinib 4 mg or 2 mg, at randomization were receiving IP and had not used high-potency TCS in the previous 14 days were enrolled in the RWDT substudy.) | 70 (At Week 52: Participants who received Baricitinib 4 mg, 2 mg, 1 mg or placebo in treatment period 1 and were not eligible for the RWDT substudy remained on their current dose of Baricitinib.) | 32 (At Week 52: Participants who received Baricitinib 4 mg, 2 mg, 1 mg or placebo in treatment period 1 and were not eligible for the RWDT substudy remained on their current dose of Baricitinib.) | 249 (At Week 52: Participants who received Baricitinib 4 mg, 2 mg, 1 mg or placebo in treatment period 1 and were not eligible for the RWDT substudy remained on their current dose of Baricitinib.) | 264 (At Week 52: Participants who received Baricitinib 4 mg, 2 mg, 1 mg or placebo in treatment period 1 and were not eligible for the RWDT substudy remained on their current dose of Baricitinib.)
Received at Least 1 Dose of IP | 0 | 0 | 0 | 0 | 0 | 92 | 91 | 92 | 84 | 84 | 84 | 70 | 32 | 249 | 264
Completed (Regarding the participants who did not complete the study due to the reason "study termination by sponsor". As pre-planned in the protocol, study termination may have occurred in a specific country or region when baricitinib was approved for the treatment of AD and became reimbursed or commercially available in that country or region, or a negative regulatory opinion was received in that country or region.) | 0 | 0 | 0 | 0 | 0 | 29 | 40 | 38 | 34 | 40 | 35 | 28 | 23 | 60 | 68
Not Completed | 0 | 0 | 0 | 0 | 0 | 63 | 51 | 54 | 50 | 44 | 49 | 42 | 9 | 189 | 196
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 17 | 21 | 17 | 19 | 15 | 17 | 16 | 3 | 66 | 70
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 13 | 10 | 11 | 7 | 12 | 8 | 7 | 2 | 63 | 72
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 23 | 15 | 20 | 17 | 10 | 11 | 8 | 0 | 41 | 32
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 2 | 2 | 3 | 9 | 3 | 2 | 11 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 1 | 1 | 1 | 0 | 4 | 4
Not completed — Withdrawal due to Caregiver Circumstances | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician is retiring | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat Population: All participants who received at least one dose of investigational product (IP) in JAHN.
Groups:
- Bari 1-mg: Participants from previous Baricitinib monotherapy studies (JAHL, JAHM) were randomized or assigned to this arm to receive Baricitinib 1 mg orally.
- Total: Total of all reporting groups
Arm/Group | Placebo | Bari 1-mg | Bari 2-mg | Bari 4-mg | Bari 2-mg Open-Label Addendum | Total
Number analyzed (Participants) | 91 | 45 | 519 | 743 | 247 | 1645
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (14.06) | 33.5 (8.49) | 34.2 (12.69) | 35.6 (12.85) | 34.9 (12.98) | 34.9 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 16 | 206 | 239 | 112 | 617
  Male | 47 | 29 | 313 | 504 | 135 | 1028
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 10 | 70 | 87 | 72 | 254
  Not Hispanic or Latino | 57 | 32 | 332 | 467 | 165 | 1053
  Unknown or Not Reported | 19 | 3 | 117 | 189 | 10 | 338
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 4 | 10 | 6 | 16 | 42
  Asian | 32 | 7 | 174 | 282 | 13 | 508
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 1 | 1 | 3
  White | 48 | 32 | 315 | 429 | 211 | 1035
  More than one race | 5 | 2 | 18 | 23 | 6 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 6 | 2 | 36 | 46 | 24 | 114
  Hungary | 7 | 2 | 15 | 21 | 27 | 72
  Czechia | 3 | 3 | 22 | 46 | 28 | 102
  Japan | 11 | 3 | 89 | 141 | 0 | 244
  Switzerland | 0 | 1 | 5 | 9 | 3 | 18
  India | 5 | 0 | 7 | 19 | 0 | 31
  Spain | 2 | 1 | 27 | 26 | 24 | 80
  Russia | 0 | 1 | 9 | 13 | 28 | 51
  Austria | 2 | 0 | 12 | 23 | 12 | 49
  South Korea | 9 | 1 | 39 | 58 | 0 | 107
  Taiwan | 8 | 2 | 30 | 50 | 0 | 90
  Denmark | 0 | 0 | 0 | 0 | 7 | 7
  Poland | 10 | 7 | 45 | 70 | 0 | 132
  Italy | 7 | 4 | 16 | 26 | 15 | 68
  Mexico | 9 | 5 | 29 | 21 | 43 | 107
  Israel | 1 | 0 | 16 | 13 | 4 | 34
  France | 0 | 0 | 15 | 19 | 0 | 34
  Australia | 4 | 1 | 30 | 42 | 32 | 109
  Germany | 7 | 12 | 77 | 100 | 0 | 196

OUTCOME MEASURES:

1. Primary Outcome: Responder and Partial Responders (RPR): Percentage of Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved a Response of Investigator's Global Assessment (IGA) 0 or 1
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
  The results were analyzed using non-responder imputation (NRI). All participants who either discontinued the study treatment or discontinued the study for any reason at any time were defined as non-responders for the NRI analysis for categorical variables such as IGA 0/1.
Time Frame: Weeks 16, 36 and 52
Population: Modified Intent-to-treat Population: All RPR participants who received at least one dose of IP in JAHN. The participants here are from the previous Baricitinib monotherapy studies (JAHL and JAHM) as the results are presented as subsets of overall RPR population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RPR-Placebo: RPR participants from previous Baricitinib monotherapy studies-JAHL and JAHM were assigned to remain in this arm to receive placebo orally.
- RPR-Bari 1-mg: RPR participants from previous Baricitinib monotherapy studies-JAHL and JAHM were assigned to remain in this arm to receive Baricitinib 1 mg orally.
- RPR-Bari 2-mg: RPR participants from previous Baricitinib monotherapy studies-JAHL and JAHM were assigned to remain in this arm to receive Baricitinib 2 mg orally.
- RPR-Bari 4-mg: RPR participants from previous Baricitinib monotherapy studies-JAHL and JAHM were assigned to remain in this arm to receive Baricitinib 4 mg orally.
Arm/Group | RPR-Placebo | RPR-Bari 1-mg | RPR-Bari 2-mg | RPR-Bari 4-mg
Number analyzed (Participants) | 52 | 45 | 54 | 70
Percentage of participants
  Week 16 | 36.5 [24.8 to 50.1] | 46.7 [32.9 to 60.9] | 59.3 [46.0 to 71.3] | 48.6 [37.2 to 60.0]
  Week 36 | 23.1 [13.7 to 36.1] | 31.1 [19.5 to 45.7] | 63.0 [49.6 to 74.6] | 37.1 [26.8 to 48.9]
  Week 52 | 28.8 [18.3 to 42.3] | 35.6 [23.2 to 50.2] | 50.0 [37.1 to 62.9] | 40.0 [29.3 to 51.7]

2. Primary Outcome: RPR: Percentage of Participants From Combination Therapy Study (JAIY) Who Achieved a Response of IGA 0 or 1
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
  The results were analyzed using NRI. All participants who either discontinued the study treatment or discontinued the study for any reason at any time were defined as non-responders for the NRI analysis for categorical variables such as IGA 0/1.
Time Frame: Weeks 16, 36, and 52
Population: Modified Intent-to-treat Population: All RPR participants who received at least one dose of IP in JAHN. The participants here are from the previous Baricitinib combination therapy study (JAIY) as the results are presented as subsets of overall RPR population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RPR-Placebo: RPR participants from previous Baricitinib combination therapy study-JAIY were assigned to remain in this arm to receive placebo orally.
- RPR-Bari 2-mg: RPR participants from previous Baricitinib combination therapy study-JAIY were assigned to remain in this arm to receive Baricitinib 2 mg orally.
- RPR-Bari 4-mg: RPR participants from previous Baricitinib combination therapy study JAIY were assigned to remain in this arm to receive Baricitinib 4 mg orally.
Arm/Group | RPR-Placebo | RPR-Bari 2-mg | RPR-Bari 4-mg
Number analyzed (Participants) | 34 | 53 | 63
Percentage of participants
  Week 16 | 47.1 [31.5 to 63.3] | 45.3 [32.7 to 58.5] | 31.7 [21.6 to 44.0]
  Week 36 | 41.2 [26.4 to 57.8] | 24.5 [14.9 to 37.6] | 30.2 [20.2 to 42.4]
  Week 52 | 29.4 [16.8 to 46.2] | 30.2 [19.5 to 43.5] | 31.7 [21.6 to 44.0]

3. Secondary Outcome: RPR: Percentage of Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved a Response of IGA 0, 1 or 2
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
  The results were analyzed using NRI. All participants who either discontinued the study treatment or discontinued the study for any reason at any time were defined as non-responders for the NRI analysis for categorical variables such as IGA 0/1/2.
Time Frame: Weeks 16, 36, and 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RPR-Placebo | RPR-Bari 1-mg | RPR-Bari 2-mg | RPR-Bari 4-mg
Number analyzed (Participants) | 52 | 45 | 54 | 70
Percentage of participants
  Week 16 | 69.2 [55.7 to 80.1] | 77.8 [63.7 to 87.5] | 81.5 [69.2 to 89.6] | 72.9 [61.5 to 81.9]
  Week 36 | 48.1 [35.1 to 61.3] | 60.0 [45.5 to 73.0] | 81.5 [69.2 to 89.6] | 58.6 [46.9 to 69.4]
  Week 52 | 46.2 [33.3 to 59.5] | 53.3 [39.1 to 67.1] | 72.2 [59.1 to 82.4] | 58.6 [46.9 to 69.4]

4. Secondary Outcome: RPR: Percentage of Participants From Combination Therapy Study (JAIY) Who Achieved a Response of IGA 0, 1, or 2
Description: as for outcome 3
Time Frame: Weeks 16, 36, and 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RPR Placebo: RPR participants from previous Baricitinib combination therapy study-JAIY were assigned to remain in this arm to receive placebo orally.
- RPR Bari 2 mg: RPR participants from previous Baricitinib combination therapy study-JAIY were assigned to remain in this arm to receive Baricitinib 2 mg orally.
- RPR Bari 4 mg: RPR participants from previous Baricitinib combination therapy study-JAIY were assigned to remain in this arm to receive Baricitinib 4 mg orally.
Arm/Group | RPR Placebo | RPR Bari 2 mg | RPR Bari 4 mg
Number analyzed (Participants) | 34 | 53 | 63
Percentage of participants
  Week 16 | 70.6 [53.8 to 83.2] | 73.6 [60.4 to 83.6] | 63.5 [51.1 to 74.3]
  Week 36 | 55.9 [39.5 to 71.1] | 49.1 [36.1 to 62.1] | 52.4 [40.3 to 64.2]
  Week 52 | 50.0 [34.1 to 65.9] | 54.7 [41.5 to 67.3] | 52.4 [40.3 to 64.2]

5. Secondary Outcome: Non Responders (NR): Percentage of Baricitinib NR Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved a Response of IGA 0, 1 or 2
Description: as for outcome 3
Time Frame: Weeks 16, 36 and 52
Population: Modified Intent-to-treat Population: All NR participants who received at least one dose of IP in JAHN. The participants here are from previous the Baricitinib monotherapy studies (JAHL and JAHM) as the results are presented as subsets of overall NR population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- NR: Bari 1 mg to 2 mg: NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM who received Baricitinib 1 mg and were re-randomized to this arm to receive Baricitinib 2 mg orally.
- NR: Bari 2 mg to 2 mg: NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM who received Baricitinib 2 mg and were re-randomized to this arm to receive Baricitinib 2 mg orally.
- NR: Bari 2 mg to 4 mg: NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM who received Baricitinib 2 mg and were re-randomized to this arm to receive Baricitinib 4 mg orally.
- NR: Bari 4 mg to 4 mg: NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM who received Baricitinib 4 mg and were re-randomized to this arm to receive Baricitinib 4 mg orally.
Arm/Group | NR: Bari 1 mg to 2 mg | NR: Bari 1 mg to 4 mg | NR: Bari 2 mg to 2 mg | NR: Bari 2 mg to 4 mg | NR: Bari 4 mg to 4 mg
Number analyzed (Participants) | 87 | 81 | 84 | 78 | 156
Percentage of participants
  Week 16 | 46.0 [35.9 to 56.4] | 55.6 [44.7 to 65.9] | 47.6 [37.3 to 58.2] | 43.6 [33.1 to 54.6] | 40.4 [33.0 to 48.2]
  Week 36 | 40.2 [30.6 to 50.7] | 43.2 [33.0 to 54.1] | 44.0 [33.9 to 54.7] | 48.7 [37.9 to 59.6] | 39.1 [31.8 to 46.9]
  Week 52 | 31.0 [22.3 to 41.4] | 48.1 [37.6 to 58.9] | 44.0 [33.9 to 54.7] | 38.5 [28.4 to 49.6] | 41.0 [33.6 to 48.9]

6. Secondary Outcome: NR: Percentage of Baricitinib NR Participants From Combination Therapy Study (JAIY) Who Achieved a Response of IGA 0, 1 or 2
Description: as for outcome 3
Time Frame: Weeks 16, 36, and 52
Population: Modified Intent-to-treat Population: All NR participants who received at least one dose of IP in JAHN. The participants here are from previous the previous Baricitinib combination therapy study (JAIY) as the results are presented as subsets of overall NR population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- NR: Bari 2 mg to 2 mg: NR participants from previous Baricitinib combination therapy study-JAIY who received Baricitinib 2 mg and were re-randomized to this arm to receive Baricitinib 2 mg orally.
- NR: Bari 2 mg to 4 mg: NR participants from previous Baricitinib combination therapy study-JAIY who received Baricitinib 2 mg and were re-randomized to this arm to receive Baricitinib 4 mg orally.
- NR: Bari 4 mg to 4 mg: NR participants from previous Baricitinib combination therapy study-JAIY who received Baricitinib 4 mg and were re-randomized to this arm to receive Baricitinib 4 mg orally.
Arm/Group | NR: Bari 2 mg to 2 mg | NR: Bari 2 mg to 4 mg | NR: Bari 4 mg to 4 mg
Number analyzed (Participants) | 20 | 21 | 39
Percentage of participants
  Week 16 | 35.0 [18.1 to 56.7] | 57.1 [36.5 to 75.5] | 30.8 [18.6 to 46.4]
  Week 36 | 40.0 [21.9 to 61.3] | 42.9 [24.5 to 63.5] | 20.5 [10.8 to 35.5]
  Week 52 | 45.0 [25.8 to 65.8] | 42.9 [24.5 to 63.5] | 28.2 [16.5 to 43.8]

7. Secondary Outcome: NR: Percentage of Baricitinib NR Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved a Response of IGA 0 or 1
Description: as for outcome 2
Time Frame: Weeks 16, 36, 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Bari 1 mg to 2 mg | NR: Bari 1 mg to 4 mg | NR: Bari 2 mg to 2 mg | NR: Bari 2 mg to 4 mg | NR: Bari 4 mg to 4 mg
Number analyzed (Participants) | 87 | 81 | 84 | 78 | 156
Percentage of participants
  Week 16 | 13.8 [8.1 to 22.6] | 23.5 [15.6 to 33.8] | 15.5 [9.3 to 24.7] | 17.9 [11.0 to 27.9] | 10.3 [6.4 to 16.0]
  Week 36 | 13.8 [8.1 to 22.6] | 12.3 [6.8 to 21.3] | 10.7 [5.7 to 19.1] | 16.7 [10.0 to 26.5] | 16.7 [11.6 to 23.3]
  Week 52 | 12.6 [7.2 to 21.2] | 12.3 [6.8 to 21.3] | 19.0 [12.1 to 28.7] | 15.4 [9.0 to 25.0] | 20.5 [14.9 to 27.5]

8. Secondary Outcome: NR: Percentage of Baricitinib NR Participants From Combination Therapy Study (JAIY) Who Achieved a Response of IGA 0 or 1
Description: as for outcome 2
Time Frame: Weeks 16, 36, and 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Bari 2 mg to 2 mg | NR: Bari 2 mg to 4 mg | NR: Bari 4 mg to 4 mg
Number analyzed (Participants) | 20 | 21 | 39
Percentage of participants
  Week 16 | 10.0 [2.8 to 30.1] | 28.6 [13.8 to 50.0] | 5.1 [1.4 to 16.9]
  Week 36 | 15.0 [5.2 to 36.0] | 23.8 [10.6 to 45.1] | 15.4 [7.2 to 29.7]
  Week 52 | 15.0 [5.2 to 36.0] | 19.0 [7.7 to 40.0] | 5.1 [1.4 to 16.9]

9. Secondary Outcome: RPR: Percentage of Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved a Response of Eczema Area and Severity Index (EASI)75
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (no disease) to 72 (severe disease). The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score.
  The results were analyzed using NRI. All participants who either discontinued the study treatment or discontinued the study for any reason at any time were defined as non-responders for the NRI analysis for categorical variables such as EASI 75.
Time Frame: Weeks 16, 36, and 52 Weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RPR-Placebo: RPR participants from previous Baricitinib monotherapy studies-JAHL and JAHM were randomized were assigned to remain in this arm to receive placebo orally.
Arm/Group | RPR-Placebo | RPR-Bari 1-mg | RPR-Bari 2-mg | RPR-Bari 4-mg
Number analyzed (Participants) | 52 | 45 | 54 | 70
Percentage of participants
  Week 16 | 42.3 [29.9 to 55.8] | 62.2 [47.6 to 74.9] | 70.4 [57.2 to 80.9] | 64.3 [52.6 to 74.5]
  Week 36 | 44.2 [31.6 to 57.7] | 46.7 [32.9 to 60.9] | 74.1 [61.1 to 83.9] | 51.4 [40.0 to 62.8]
  Week 52 | 38.5 [26.5 to 52.0] | 51.1 [37.0 to 65.0] | 64.8 [51.5 to 76.2] | 51.4 [40.0 to 62.8]

10. Secondary Outcome: RPR: Percentage of Participants From Combination Therapy Study (JAIY) Who Achieved a Response of EASI 75
Description: as for outcome 9
Time Frame: Weeks 16, 36, and 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RPR-Bari 4-mg: RPR participants from previous Baricitinib combination therapy study-JAIY were assigned to remain in this arm to receive Baricitinib 4 mg orally.
Arm/Group | RPR-Placebo | RPR-Bari 2-mg | RPR-Bari 4-mg
Number analyzed (Participants) | 34 | 53 | 63
Percentage of participants
  Week 16 | 55.9 [39.5 to 71.1] | 67.9 [54.5 to 78.9] | 55.6 [43.3 to 67.2]
  Week 36 | 47.1 [31.5 to 63.3] | 47.2 [34.4 to 60.3] | 44.4 [32.8 to 56.7]
  Week 52 | 38.2 [23.9 to 55.0] | 52.8 [39.7 to 65.6] | 42.9 [31.4 to 55.1]

11. Secondary Outcome: NR: Percentage of Baricitinib NR Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved a Response of EASI 75
Description: as for outcome 9
Time Frame: Weeks 16, 36, and 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Bari 1 mg to 2 mg | NR: Bari 1 mg to 4 mg | NR: Bari 2 mg to 2 mg | NR: Bari 2 mg to 4 mg | NR: Bari 4 mg to 4 mg
Number analyzed (Participants) | 87 | 81 | 84 | 78 | 156
Percentage of participants
  Week 16 | 33.3 [24.3 to 43.8] | 43.2 [33.0 to 54.1] | 38.1 [28.4 to 48.8] | 38.5 [28.4 to 49.6] | 26.9 [20.6 to 34.4]
  Week 36 | 32.2 [23.3 to 42.6] | 30.9 [21.9 to 41.6] | 31.0 [22.1 to 41.5] | 44.9 [34.3 to 55.9] | 30.8 [24.1 to 38.4]
  Week 52 | 28.7 [20.3 to 39.0] | 35.8 [26.2 to 46.7] | 34.5 [25.2 to 45.2] | 34.6 [25.0 to 45.7] | 33.3 [26.4 to 41.1]

12. Secondary Outcome: NR: Percentage of Baricitinib NR Participants From Combination Therapy Study (JAIY) Who Achieved a Response of EASI 75
Description: as for outcome 9
Time Frame: Weeks 16, 36, and 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Bari 2 mg to 2 mg | NR: Bari 2 mg to 4 mg | NR: Bari 4 mg to 4 mg
Number analyzed (Participants) | 20 | 21 | 39
Percentage of participants
  Week 16 | 20.0 [8.1 to 41.6] | 57.1 [36.5 to 75.5] | 28.2 [16.5 to 43.8]
  Week 36 | 25.0 [11.2 to 46.9] | 28.6 [13.8 to 50.0] | 23.1 [12.6 to 38.3]
  Week 52 | 20.0 [8.1 to 41.6] | 28.6 [13.8 to 50.0] | 28.2 [16.5 to 43.8]

13. Secondary Outcome: RPR: Percentage of Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved 4-Point Improvement in Itch Numeric Rating Scale (NRS)
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participants itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours. The results were analyzed using NRI. All participants who either discontinued the study treatment or discontinued the study for any reason at any time were defined as non-responders for the NRI analysis for categorical variables such as NRS.
Time Frame: Week 16
Population: Modified Intent-to-treat Population: All RPR participants who received at least one dose of IP in JAHN with Baseline Itch NRS Score >= 4. The participants here are from the previous Baricitinib monotherapy studies (JAHL and JAHM) as the results are presented as subsets of overall RPR population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RPR-Placebo | RPR-Bari 1-mg | RPR-Bari 2-mg | RPR-Bari 4-mg
Number analyzed (Participants) | 43 | 31 | 43 | 61
Percentage of participants | 32.6 [20.5 to 47.5] | 25.8 [13.7 to 43.2] | 32.6 [20.5 to 47.5] | 41.0 [29.5 to 53.5]

14. Secondary Outcome: RPR: Percentage of Participants From Combination Therapy Study (JAIY) Who Achieved 4-Point Improvement in Itch NRS
Description: as for outcome 13
Time Frame: Week 16
Population: Modified Intent-to-treat Population: All RPR participants who received at least one dose of IP in JAHN with Baseline Itch NRS Score >= 4. The participants here are from the previous Baricitinib combination therapy study (JAIY) as the results are presented as subsets of overall RPR population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RPR Placebo | RPR Bari 2 mg | RPR Bari 4 mg
Number analyzed (Participants) | 32 | 48 | 56
Percentage of participants | 37.5 [22.9 to 54.7] | 45.8 [32.6 to 59.7] | 46.4 [34.0 to 59.3]

15. Secondary Outcome: NR: Percentage of Baricitinib NR Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved 4-Point Improvement in Itch NRS
Description: as for outcome 13
Time Frame: Week 16
Population: Modified Intent-to-treat Population: All NR participants who received at least one dose of IP in JAHN with Baseline Itch NRS Score >= 4. The participants here are from previous the Baricitinib monotherapy studies (JAHL and JAHM) as the results are presented as subsets of overall NR population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Bari 1 mg to 2 mg | NR: Bari 1 mg to 4 mg | NR: Bari 2 mg to 2 mg | NR: Bari 2 mg to 4 mg | NR: Bari 4 mg to 4 mg
Number analyzed (Participants) | 80 | 62 | 70 | 71 | 138
Percentage of participants | 20.0 [12.7 to 30.0] | 38.7 [27.6 to 51.2] | 24.3 [15.8 to 35.5] | 31.0 [21.4 to 42.5] | 22.5 [16.3 to 30.1]

16. Secondary Outcome: NR: Percentage of Baricitinib NR Participants From Combination Therapy Study (JAIY) Who Achieved 4-Point Improvement in Itch NRS
Description: as for outcome 13
Time Frame: Week 16
Population: Modified Intent-to-treat Population: All NR participants who received at least one dose of IP in JAHN with Baseline Itch NRS Score >= 4. The participants here are from previous the previous Baricitinib combination therapy study (JAIY) as the results are presented as subsets of overall NR population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Bari 2 mg to 2 mg | NR: Bari 2 mg to 4 mg | NR: Bari 4 mg to 4 mg
Number analyzed (Participants) | 19 | 19 | 35
Percentage of participants | 31.6 [15.4 to 54.0] | 36.8 [19.1 to 59.0] | 31.4 [18.6 to 48.0]

17. Secondary Outcome: NR: Percentage of Placebo NR Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved a Response of IGA 0, 1 or 2
Description: as for outcome 3
Time Frame: Weeks 4, 16, 24, 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- NR: Placebo to Bari 2 mg: NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM who received placebo and were re-randomized to this arm to receive Baricitinib 2 mg orally.
- NR: Placebo to Bari 4 mg: NR participants from previous Baricitinib monotherapy studies-JAHL and JAHM who received placebo and were re-randomized to this arm to receive Baricitinib 4 mg orally.
Arm/Group | NR: Placebo to Bari 2 mg | NR: Placebo to Bari 4 mg
Number analyzed (Participants) | 180 | 194
Percentage of participants
  Week 4 | 57.8 [50.5 to 64.8] | 67.0 [60.1 to 73.2]
  Week 16 | 56.7 [49.4 to 63.7] | 62.9 [55.9 to 69.4]
  Week 24 | 55.6 [48.3 to 62.6] | 57.2 [50.2 to 64.0]
  Week 52 | 50.6 [43.3 to 57.8] | 46.9 [40.0 to 53.9]

18. Secondary Outcome: NR: Percentage of Placebo NR Participants From Combination Therapy Study (JAIY) Who Achieved a Response of IGA 0, 1 or 2
Description: as for outcome 3
Time Frame: Weeks 4, 16, 24, 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- NR: Placebo to Bari 2 mg: NR participants from previous Baricitinib combination therapy study-JAIY who received placebo and were re-randomized to this arm to receive Baricitinib 2 mg orally.
- NR: Placebo to Bari 4 mg: NR participants from previous Baricitinib combination therapy study-JAIY who received placebo and were re-randomized to this arm to receive Baricitinib 4 mg orally.
Arm/Group | NR: Placebo to Bari 2 mg | NR: Placebo to Bari 4 mg
Number analyzed (Participants) | 34 | 28
Percentage of participants
  Week 4 | 50.0 [34.1 to 65.9] | 46.4 [29.5 to 64.2]
  Week 16 | 47.1 [31.5 to 63.3] | 46.4 [29.5 to 64.2]
  Week 24 | 38.2 [23.9 to 55.0] | 39.3 [23.6 to 57.6]
  Week 52 | 26.5 [14.6 to 43.1] | 25.0 [12.7 to 43.4]

19. Secondary Outcome: NR: Percentage of Placebo NR Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved a Response of IGA 0 or 1
Description: as for outcome 2
Time Frame: Weeks 4, 16, 24, 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Placebo to Bari 2 mg | NR: Placebo to Bari 4 mg
Number analyzed (Participants) | 180 | 194
Percentage of participants
  Week 4 | 22.8 [17.3 to 29.4] | 25.8 [20.1 to 32.4]
  Week 16 | 22.2 [16.8 to 28.8] | 29.9 [23.9 to 36.7]
  Week 24 | 22.2 [16.8 to 28.8] | 27.8 [22.0 to 34.5]
  Week 52 | 20.6 [15.3 to 27.0] | 23.7 [18.3 to 30.2]

20. Secondary Outcome: NR: Percentage of Placebo NR Participants From Combination Therapy Study (JAIY) Who Achieved a Response of IGA 0 or 1
Description: as for outcome 2
Time Frame: Weeks 4, 16, 24, 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Placebo to Bari 2 mg | NR: Placebo to Bari 4 mg
Number analyzed (Participants) | 34 | 28
Percentage of participants
  Week 4 | 0 [0.0 to 10.2] | 14.3 [5.7 to 31.5]
  Week 16 | 5.9 [1.6 to 19.1] | 25.0 [12.7 to 43.4]
  Week 24 | 11.8 [4.7 to 26.6] | 17.9 [7.9 to 35.6]
  Week 52 | 5.9 [1.6 to 19.1] | 10.7 [3.7 to 27.2]

21. Secondary Outcome: NR: Percentage of Placebo NR Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved a Response of EASI 75
Description: as for outcome 9
Time Frame: Weeks 4, 16, 24, 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Placebo to Bari 2 mg | NR: Placebo to Bari 4 mg
Number analyzed (Participants) | 180 | 194
Percentage of participants
  Week 4 | 38.9 [32.1 to 46.2] | 46.9 [40.0 to 53.9]
  Week 16 | 43.9 [36.8 to 51.2] | 53.6 [46.6 to 60.5]
  Week 24 | 45.0 [37.9 to 52.3] | 45.4 [38.5 to 52.4]
  Week 52 | 41.1 [34.2 to 48.4] | 38.7 [32.1 to 45.7]

22. Secondary Outcome: NR: Percentage of Placebo NR Participants From Combination Therapy Study (JAIY) Who Achieved a Response of EASI 75
Description: as for outcome 9
Time Frame: Weeks 4, 16, 24, 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Placebo to Bari 2 mg | NR: Placebo to Bari 4 mg
Number analyzed (Participants) | 34 | 28
Percentage of participants
  Week 4 | 23.5 [12.4 to 40.0] | 39.3 [23.6 to 57.6]
  Week 16 | 38.2 [23.9 to 55.0] | 39.3 [23.6 to 57.6]
  Week 24 | 32.4 [19.1 to 49.2] | 32.1 [17.9 to 50.7]
  Week 52 | 26.5 [14.6 to 43.1] | 32.1 [17.9 to 50.7]

23. Secondary Outcome: NR: Percentage of Placebo NR Participants From Monotherapy Studies (JAHL, JAHM) Who Achieved 4-Point Improvement in Itch NRS
Description: as for outcome 13
Time Frame: Week 16
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Placebo to Bari 2 mg | NR: Placebo to Bari 4 mg
Number analyzed (Participants) | 165 | 171
Percentage of participants | 33.9 [27.2 to 41.5] | 35.7 [28.9 to 43.1]

24. Secondary Outcome: NR: Percentage of Placebo NR Participants From Combination Therapy Study (JAIY) Who Achieved 4-Point Improvement in Itch NRS
Description: as for outcome 13
Time Frame: Week 16
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NR: Placebo to Bari 2 mg | NR: Placebo to Bari 4 mg
Number analyzed (Participants) | 34 | 26
Percentage of participants | 20.6 [10.3 to 36.8] | 26.9 [13.7 to 46.1]

25. Secondary Outcome: Percentage of Participants Who Achieved a Response of IGA 0, 1, or 2 Assessed at 16 Weeks After Rerandomization (Week 68) and Week 104 in Randomized Withdrawal and Downtitration Substudy (Participants Entering the Substudy)
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification. All missing values were imputed using modified last observation carried forward (mLOCF).
Time Frame: Weeks 68, 104
Population: Randomized Downtitration Withdrawal Substudy Population: All participants (including open-label participants) who are rerandomized at Week 52, entered the substudy, and received at least 1 dose of the IP in Period 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 2 mg Bari to 2 mg Bari Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to Placebo Substudy
Number analyzed (Participants) | 84 | 84 | 84 | 92 | 91 | 92
Percentage of participants
  Week 68 | 86.9 [78.1 to 92.5] | 60.7 [50.0 to 70.5] | 50.0 [39.5 to 60.5] | 92.4 [85.1 to 96.3] | 70.3 [60.3 to 78.7] | 44.6 [34.8 to 54.7]
  Week 104 | 85.7 [76.7 to 91.6] | 48.8 [38.4 to 59.3] | 41.7 [31.7 to 52.3] | 83.7 [74.8 to 89.9] | 58.2 [48.0 to 67.8] | 33.7 [24.9 to 43.8]

26. Secondary Outcome: Percentage of Participants Who Achieved a Response of IGA 0 or 1 Assessed at 16 Weeks After Rerandomization (Week 68) and Week 104 in Randomized Withdrawal and Downtitration Substudy (Participants Entering the Substudy)
Description: as for outcome 25
Time Frame: Weeks 68, 104
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 2 mg Bari to 2 mg Bari Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to Placebo Substudy
Number analyzed (Participants) | 84 | 84 | 84 | 92 | 91 | 92
Percentage of participants
  Week 68 | 51.2 [40.7 to 61.6] | 45.2 [35.0 to 55.9] | 29.8 [21.0 to 40.2] | 47.8 [37.9 to 57.9] | 41.8 [32.2 to 52.0] | 25.0 [17.3 to 34.7]
  Week 104 | 47.6 [37.3 to 58.2] | 35.7 [26.3 to 46.4] | 33.3 [24.2 to 43.9] | 42.4 [32.8 to 52.6] | 38.5 [29.1 to 48.7] | 21.7 [14.5 to 31.2]

27. Secondary Outcome: Percentage of Participants Achieving Response of EASI75 From Baseline of Originating Study Assessed at 16 Weeks After Rerandomization (Week 68) and Week 104 in Randomized Withdrawal and Downtitration Substudy (Participants Entering the Substudy)
Description: as for outcome 9
Time Frame: Weeks 68, 104
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 2 mg Bari to 2 mg Bari Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to Placebo Substudy
Number analyzed (Participants) | 84 | 84 | 84 | 92 | 91 | 92
Percentage of participants
  Week 68 | 79.8 [70.0 to 87.0] | 58.3 [47.7 to 68.3] | 45.2 [35.0 to 55.9] | 73.9 [64.1 to 81.8] | 69.2 [59.1 to 77.8] | 44.6 [34.8 to 54.7]
  Week 104 | 73.8 [63.5 to 82.0] | 58.3 [47.7 to 68.3] | 41.7 [31.7 to 52.3] | 72.8 [63.0 to 80.9] | 58.2 [48.0 to 67.8] | 43.5 [33.8 to 53.7]

28. Secondary Outcome: Time to Retreatment (Time to IGA ≥3) in Randomized Withdrawal and Down Titration (Participants Entering the Sub Study)
Description: Participants who entered the Substudy, relapsed with an IGA ≥3 and were retreated
Time Frame: Week 52 Up to Week 200
Population: Participants who received at least one dose of study medication during Week 52 to Week 200 in Study JAHN, entered the randomized down titration withdrawal sub study, relapsed with an IGA ≥3 and were retreated from Week 52 up to Week 200.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 4 mg Bari to 4 mg Bari Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 2 mg Bari to 2 mg Bari Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to Placebo Substudy
Number analyzed (Participants) | 39 | 47 | 50 | 49 | 45 | 63
Days | 117.0 [57.0 to 289.0] | 56.0 [29.0 to 170.0] | 29.5 [26.0 to 113.0] | 61.0 [29.0 to 269.0] | 169.0 [56.0 to 368.0] | 30.0 [28.0 to 87.0]

29. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1, or 2 Assessed at 16 Weeks After Rerandomization (Week 68) and Week 104 in Randomized Withdrawal and Downtitration Substudy (Participants Entering the Substudy With IGA 0 or 1)
Description: as for outcome 25
Time Frame: Weeks 68, 104
Population: Randomized Downtitration Withdrawal Substudy Population with Week 52 IGA of 0 or 1: All participants (including open-label participants) who are rerandomized at Week 52, entered the substudy with IGA 0 or 1, and received atleast 1 dose of the IP in Period 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 2 mg Bari to 2 mg Bari Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to Placebo Substudy
Number analyzed (Participants) | 43 | 43 | 43 | 48 | 48 | 49
Percentage of participants
  Week 68 | 97.7 [87.9 to 99.6] | 76.7 [62.3 to 86.8] | 72.1 [57.3 to 83.3] | 95.8 [86.0 to 98.8] | 89.6 [77.8 to 95.5] | 55.1 [41.3 to 68.1]
  Week 104 | 90.7 [78.4 to 96.3] | 69.8 [54.9 to 81.4] | 62.8 [47.9 to 75.6] | 93.8 [83.2 to 97.9] | 77.1 [63.5 to 86.7] | 42.9 [30.0 to 56.7]

30. Secondary Outcome: Percentage of Participants With a Response of IGA 0 or 1 Assessed at 16 Weeks After Rerandomization (Week 68) and Week 104 in Randomized Withdrawal and Downtitration Substudy (Participants Entering the Substudy With IGA 0 or 1)
Description: as for outcome 25
Time Frame: Weeks 68, 104
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 2 mg Bari to 2 mg Bari Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to Placebo Substudy
Number analyzed (Participants) | 43 | 43 | 43 | 48 | 48 | 49
Percentage of participants
  Week 68 | 74.4 [59.8 to 85.1] | 69.8 [54.9 to 81.4] | 55.8 [41.1 to 69.6] | 70.8 [56.8 to 81.8] | 66.7 [52.5 to 78.3] | 36.7 [24.7 to 50.7]
  Week 104 | 62.8 [47.9 to 75.6] | 55.8 [41.1 to 69.6] | 58.1 [43.3 to 71.6] | 60.4 [46.3 to 73.0] | 60.4 [46.3 to 73.0] | 32.7 [21.2 to 46.6]

31. Secondary Outcome: Percentage of Participants With a Response of EASI75 From Baseline of Originating Study Assessed at 16 Weeks After Rerandomization(Week 68) and Week 104 in Randomized Withdrawal and Downtitration Substudy (Participants Entering Substudy With IGA 0 or 1)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 (no disease) to 72 (severe disease). The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Weeks 68, 104
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 2 mg Bari to 2 mg Bari Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to Placebo Substudy
Number analyzed (Participants) | 43 | 43 | 43 | 48 | 48 | 49
Percentage of participants
  Week 68 | 93 [81.4 to 97.6] | 76.7 [62.3 to 86.8] | 72.1 [57.3 to 83.3] | 83.3 [70.4 to 91.3] | 89.6 [77.8 to 95.5] | 63.3 [49.3 to 75.3]
  Week 104 | 76.7 [62.3 to 86.8] | 74.4 [59.8 to 85.1] | 67.4 [52.5 to 79.5] | 83.3 [70.4 to 91.3] | 79.2 [65.7 to 88.3] | 55.1 [41.3 to 68.1]

32. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1, or 2 Assessed Within 16 Weeks of Retreatment (Week 68) Randomized Withdrawal and Downtitration (Participants Retreated During Substudy)
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification. All missing values were imputed using modified last observation carried forward (mLOCF).
Time Frame: Week 68
Population: Re-Treatment Substudy Population: A subset of Randomized Downtitration Withdrawal Substudy Population who experienced IGA ≥3 at any time in Period 2 and received at least 1 dose of retreatment of the original dose.
Measure: Number; unit: Percentage of participants
Groups:
- 4 mg Bari to 4 mg Bari Substudy: Participants who received Baricitinib 4 mg at the start of Study JAHN are rerandomized at week 52 or assigned to this arm to receive Baricitinib 4 mg orally.
- 4 mg Bari to 2 mg Bari Substudy: Participants who received Baricitinib 4 mg at the start of Study JAHN are rerandomized at week 52 or assigned to this arm to receive Baricitinib 2 mg orally.
- 4 mg Bari to Placebo Substudy: Participants who received Baricitinib 4 mg at the start of Study JAHN are rerandomized at week 52 or assigned to this arm to receive placebo orally.
- 2 mg Bari to 2 mg Bari Substudy: Participants who received Baricitinib 2 mg at the start of Study JAHN are rerandomized at week 52 or assigned to this arm to receive Baricitinib 2 mg orally.
- 2 mg Bari to 1 mg Bari Substudy: Participants who received Baricitinib 2 mg at the start of Study JAHN are rerandomized at week 52 or assigned to this arm to receive Baricitinib 1 mg orally.
- 2 mg Bari to Placebo Substudy: Participants who received Baricitinib 2 mg at the start of Study JAHN are rerandomized at week 52 or assigned to this arm to receive placebo orally.
Arm/Group | 4 mg Bari to 4 mg Bari Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 2 mg Bari to 2 mg Bari Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to Placebo Substudy
Number analyzed (Participants) | 39 | 47 | 50 | 49 | 45 | 63
Percentage of participants | 69.2 | 74.5 | 80.0 | 57.1 | 55.6 | 76.2

33. Secondary Outcome: Percentage of Participants With a Response of IGA 0 or 1 Assessed Within 16 Weeks of Retreatment (Week 68) Randomized Withdrawal and Downtitration (Participants Retreated During Substudy)
Description: as for outcome 25
Time Frame: Week 68
Population: as for outcome 32
Measure: Number; unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 2 mg Bari to 2 mg Bari Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to Placebo Substudy
Number analyzed (Participants) | 39 | 47 | 50 | 49 | 45 | 63
Percentage of participants | 23.1 | 25.5 | 44.0 | 10.2 | 26.7 | 39.7

34. Secondary Outcome: Percentage of Participants Achieving Response of EASI75 From Baseline of Originating Study Assessed Within 16 Weeks of Retreatment (Week 68) Randomized Withdrawal and Downtitration (Participants Retreated During Substudy)
Description: as for outcome 31
Time Frame: Week 68
Population: as for outcome 32
Measure: Number; unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 2 mg Bari to 2 mg Bari Substudy | 2 mg Bari to 1 mg Bari SubstudY | 2 mg Bari to Placebo Substudy
Number analyzed (Participants) | 39 | 47 | 50 | 49 | 45 | 63
Percentage of participants | 61.5 | 53.2 | 70.0 | 55.1 | 44.4 | 71.4

35. Secondary Outcome: Percentage of Participants With a Response of IGA 0, 1, or 2 Assessed at Week 104 (Participants Not Entered Into Substudy)
Description: as for outcome 25
Time Frame: Week 104
Population: Period 2 Nonsubstudy Population: All participants randomized at Week 0 of main Study JAHN (excluding open-label participants) who were not eligible to enter the substudy at Week 52 and received at least 1 dose of the IP in Period 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Non-substudy | 2 mg Bari to 2 mg Bari Non-substudy | 1 mg Bari to 1 mg Bari Non-substudy | Placebo to Placebo Non-substudy
Number analyzed (Participants) | 264 | 193 | 32 | 70
Percentage of participants | 41.3 [35.5 to 47.3] | 45.6 [38.7 to 52.6] | 71.9 [54.6 to 84.4] | 51.4 [40.0 to 62.8]

36. Secondary Outcome: Percentage of Participants With a Response of IGA 0 or 1 Assessed at Week 104 (Participants Not Entered Into Substudy)
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification. The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification. All missing values were imputed using modified last observation carried forward (mLOCF).
Time Frame: Week 104
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Non-substudy | 2 mg Bari to 2 mg Bari Non-substudy | 1 mg Bari to 1 mg Bari Non-substudy | Placebo to Placebo Non-substudy
Number analyzed (Participants) | 264 | 193 | 32 | 70
Percentage of participants | 13.3 [9.7 to 17.9] | 13.5 [9.4 to 19.0] | 53.1 [36.4 to 69.1] | 40.0 [29.3 to 51.7]

37. Secondary Outcome: Percentage of Participants Achieving Response of EASI75 From Baseline of Originating Study Assessed at Week 104 (Participants Not Entered Into Substudy)
Description: as for outcome 31
Time Frame: Week 104
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 4 mg Bari to 4 mg Bari Non-substudy | 2 mg Bari to 2 mg Bari Non-substudy | 1 mg Bari to 1 mg Bari Non-substudy | Placebo to Placebo Non-substudy
Number analyzed (Participants) | 264 | 193 | 32 | 70
Percentage of participants | 39.8 [34.1 to 45.8] | 40.9 [34.2 to 48.0] | 65.6 [48.3 to 79.6] | 54.3 [42.7 to 65.4]

ADVERSE EVENTS:
Time Frame: Baseline through Week 200
Description: All participants who received at least one dose of IP. The participants from open label arm were included in the Baricitinib 2-mg arm while reporting the safety data. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | Bari 1-mg | Bari 2-mg | Bari 4-mg | 2 mg Bari to Placebo Substudy | 2 mg Bari to 1 mg Bari Substudy | 2 mg Bari to 2 mg Bari Substudy | 4 mg Bari to Placebo Substudy | 4 mg Bari to 2 mg Bari Substudy | 4 mg Bari to 4 mg Bari Substudy | Placebo to Placebo Non-substudy | 1 mg Bari to 1 mg Bari Non-substudy | 2 mg Bari to 2 mg Bari Non-substudy | 4 mg Bari to 4 mg Bari Non-substudy
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/45 | 0/766 | 1/743 | 1/92 | 0/91 | 0/92 | 0/84 | 0/84 | 0/84 | 0/70 | 0/32 | 0/249 | 1/264
Serious Adverse Events (participants affected / at risk) | 5/91 | 1/45 | 32/766 | 40/743 | 2/92 | 1/91 | 3/92 | 3/84 | 1/84 | 11/84 | 1/70 | 3/32 | 16/249 | 25/264
Other Adverse Events (participants affected / at risk) | 21/91 | 14/45 | 263/766 | 268/743 | 15/92 | 27/91 | 38/92 | 16/84 | 21/84 | 42/84 | 14/70 | 14/32 | 96/249 | 110/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=91) | Bari 1-mg (N=45) | Bari 2-mg (N=766) | Bari 4-mg (N=743) | 2 mg Bari to Placebo Substudy (N=92) | 2 mg Bari to 1 mg Bari Substudy (N=91) | 2 mg Bari to 2 mg Bari Substudy (N=92) | 4 mg Bari to Placebo Substudy (N=84) | 4 mg Bari to 2 mg Bari Substudy (N=84) | 4 mg Bari to 4 mg Bari Substudy (N=84) | Placebo to Placebo Non-substudy (N=70) | 1 mg Bari to 1 mg Bari Non-substudy (N=32) | 2 mg Bari to 2 mg Bari Non-substudy (N=249) | 4 mg Bari to 4 mg Bari Non-substudy (N=264)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematotympanum (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Retinopathy proliferative (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipeloid (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis syphilitic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocephalus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dairy intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaplastic large cell lymphoma t- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiocentric lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral t-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/47 (0) | 0/29 (0) | 0/448 (0) | 0/504 (0) | 0/48 (0) | 0/61 (0) | 0/49 (0) | 0/48 (0) | 0/54 (0) | 0/53 (0) | 0/36 (0) | 0/20 (0) | 1/159 (1) | 0/190 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/47 (0) | 0/29 (0) | 0/448 (0) | 0/504 (0) | 0/48 (0) | 0/61 (0) | 0/49 (0) | 0/48 (0) | 0/54 (0) | 0/53 (0) | 0/36 (0) | 1/20 (1) | 0/159 (0) | 0/190 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/44 (0) | 0/16 (0) | 0/318 (0) | 0/239 (0) | 0/44 (0) | 0/30 (0) | 0/43 (0) | 0/36 (0) | 0/30 (0) | 0/31 (0) | 0/34 (0) | 0/12 (0) | 0/90 (0) | 1/74 (1)
Xanthogranuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/44 (0) | 0/16 (0) | 0/318 (0) | 0/239 (0) | 0/44 (0) | 0/30 (0) | 0/43 (0) | 0/36 (0) | 0/30 (0) | 0/31 (0) | 0/34 (0) | 0/12 (0) | 1/90 (1) | 0/74 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1/44 (1) | 0/16 (0) | 0/318 (0) | 0/239 (0) | 0/44 (0) | 0/30 (0) | 0/43 (0) | 0/36 (0) | 0/30 (0) | 0/31 (0) | 0/34 (0) | 0/12 (0) | 0/90 (0) | 0/74 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 10 (13) | 9 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 5 (5)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parakeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=91) | Bari 1-mg (N=45) | Bari 2-mg (N=766) | Bari 4-mg (N=743) | 2 mg Bari to Placebo Substudy (N=92) | 2 mg Bari to 1 mg Bari Substudy (N=91) | 2 mg Bari to 2 mg Bari Substudy (N=92) | 4 mg Bari to Placebo Substudy (N=84) | 4 mg Bari to 2 mg Bari Substudy (N=84) | 4 mg Bari to 4 mg Bari Substudy (N=84) | Placebo to Placebo Non-substudy (N=70) | 1 mg Bari to 1 mg Bari Non-substudy (N=32) | 2 mg Bari to 2 mg Bari Non-substudy (N=249) | 4 mg Bari to 4 mg Bari Non-substudy (N=264)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 17 (18) | 19 (20) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 7 (7) | 4 (7)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 9 (9) | 14 (15) | 7 (8) | 4 (5) | 14 (15) | 3 (4) | 7 (7) | 33 (33) | 29 (31)
Folliculitis (Infections and infestations) | 1 (2) | 0 (0) | 19 (21) | 12 (13) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 10 (10) | 6 (6)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 13 (13) | 21 (23) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 13 (16) | 26 (27)
Nasopharyngitis (Infections and infestations) | 10 (12) | 9 (15) | 106 (140) | 122 (173) | 5 (6) | 3 (3) | 10 (14) | 6 (12) | 8 (9) | 11 (14) | 1 (1) | 1 (1) | 27 (30) | 26 (32)
Oral herpes (Infections and infestations) | 2 (3) | 0 (0) | 34 (47) | 40 (51) | 1 (2) | 0 (0) | 4 (4) | 1 (7) | 4 (5) | 2 (2) | 2 (3) | 0 (0) | 9 (14) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 43 (65) | 44 (56) | 4 (4) | 3 (5) | 3 (5) | 0 (0) | 2 (2) | 5 (7) | 1 (2) | 1 (1) | 11 (16) | 10 (18)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 20 (22) | 7 (8) | 1 (1) | 2 (2) | 2 (3) | 3 (3) | 6 (7) | 5 (8) | 1 (1) | 0 (0) | 3 (3) | 5 (9)
Vulvovaginal candidiasis (Infections and infestations) | 0/44 (0) | 0/16 (0) | 4/318 (6) | 0/239 (0) | 0/44 (0) | 2/30 (3) | 1/43 (1) | 0/36 (0) | 0/30 (0) | 1/31 (1) | 0/34 (0) | 0/12 (0) | 0/90 (0) | 0/74 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 13 (13) | 10 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 6 (6)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 12 (13) | 18 (18) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 5 (5) | 6 (6)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (7) | 1 (1) | 46 (58) | 22 (37) | 3 (3) | 4 (4) | 5 (6) | 1 (4) | 1 (1) | 2 (2) | 3 (5) | 0 (0) | 14 (15) | 10 (11)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 7 (8) | 14 (19) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 4 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol: Original Protocol (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT03334435/Prot_000.pdf
  • Study Protocol: Protocol Addendum (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT03334435/Prot_001.pdf
  • Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT03334435/SAP_003.pdf